CLINICAL TRIAL: NCT06584760
Title: Research on the Impact of Chronic Pelvic Pain on Endometriosis
Status: Not yet recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2024-152
Record Dates: First submitted 2024-08-26; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pelvic Pain; Endometriosis
Keywords: Chronic pelvic pain; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Preoperative venous blood from patients with endometriosis and pathological tissue of endometriosis removed during surgery were collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometriosis group: Patients undergoing endometriosis surgery in the gynecology department of the Fourth Affiliated Hospital of Zhejiang University School of Medicine

SUMMARY:
Chronic pelvic pain (CPP) is a common disease with multiple systems and multiple causes. In recent years, the incidence rate of CPP in women has gradually increased. It is a pain symptom that originates from pelvic organs or related structures and lasts for more than 6 months. It is closely related to gynecological diseases such as endometriosis (EMs), adenomyosis, pelvic inflammatory disease (PID), uterine leiomyoma, residual ovarian syndrome, pelvic venous congestion syndrome (PCS), etc. But its pathophysiology is very complex and still needs further exploration. Recent studies have shown that central sensitization is an important mechanism for the sustained existence of CPP.

Explore the relationship between chronic pelvic pain and its postoperative outcomes, as well as preoperative endometriosis related questionnaire surveys such as such as Endometriosis Health Profile-30 (EHP-30), Central Sensitivity Inventory (CSI), Simplified McGill Pain Questionnaire (SF-MPQ). Explore the relationship between chronic pelvic pain and its postoperative outcomes, as well as in vitro detection results such as preoperative venous blood, intraoperative pathological tissue immunohistochemistry, ELISA, transcriptome sequencing in patients with endometriosis.

DETAILED DESCRIPTION:
Conduct preoperative and postoperative endometriosis related questionnaire surveys on patients, such as Endometriosis Health Profile-30 (EHP-30), Central Sensitivity Inventory (CSI), Simplified McGill Pain Questionnaire (SF-MPQ). Follow up will be conducted 1-2 months after surgery. Preoperative venous blood from patients with endometriosis and pathological tissue of endometriosis removed during surgery were collected for in vitro testing using immunohistochemistry, ELISA, transcriptome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years old;
* Endometriosis diagnosed through previous surgery (confirmed solely by visual or histopathological examination), endometriosis discovered through imaging examination, deep infiltrating nodules discovered through palpation or imaging examination, and clinically suspected endometriosis;
* No history of migraine or tension headaches;
* No history of mental illness (such as restless leg syndrome, chronic fatigue syndrome, fibromyalgia, anxiety or panic attacks, depression).

Exclusion Criteria:

* Postmenopausal state (spontaneous or surgical);
* Previous hysterectomy and/or bilateral salpingo oophorectomy (prior to preoperative visit);
* The patient or authorizer refuses.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing endometriosis surgery in the gynecology department of the Fourth Affiliated Hospital of Zhejiang University School of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Chronic pelvic pain | Within 3 days before surgery, before leaving the hospital after surgery, postoperative discharge (6 months -3 years)
  Using Simplified McGill Pain Questionnaire (SF-MPQ) for scoring
In vitro detection results | Venous blood within 3 days before surgery; Endometriosis sample excised during surgery
  The results of immunohistochemistry, ELISA, and transcriptome sequencing of preoperative venous blood and endometrial tissue excised during surgery in patients with endometriosis

CONTACTS AND LOCATIONS:
Overall Officials: Jiannan He, Study Chair — The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, No. N1, Shopping Mall Avenue, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No